CLINICAL TRIAL: NCT05257408
Title: A Phase 3 Study of Relacorilant in Combination With Nab-Paclitaxel Versus Nab-Paclitaxel Monotherapy in Advanced, Platinum-Resistant, High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian-Tube Cancer (ROSELLA)
Brief Title: Relacorilant in Combination With Nab-Paclitaxel in Advanced, Platinum-Resistant, High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian-Tube Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-556; ROSELLA Study 556 (Other: Corcept Therapeutics); GOG-3073 (Other: Gynecologic Oncology Group); ENGOT-OV72 (Other: European Network of Gyneaecological Oncological Trial Groups); APGOT-Ov10 (Other: Asia Pacific Gyneaecological Oncological Trial Groups); LACOG 0223 (Other: Latin America Cooperative Oncology Trials Group); ANZGOG2221/2023 (Other: Australia New Zealand Oncology Group)
Record Dates: First submitted 2022-02-04; First posted 2022-02-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Neoplasm; Fallopian Tube Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — 130-nm albumin-bound paclitaxel; relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel 80 mg/m^2 with Relacorilant 150 mg (Experimental): Patients receive nab-paclitaxel 80 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle in combination with intermittent relacorilant (150 mg relacorilant once daily on the day before, the day of, and the day after nab-paclitaxel), administered orally under fed conditions. Relacorilant will not be administered on Cycle 1 Day -1.
  Interventions: Drug: Nab-paclitaxel 80 mg/m^2; Drug: Relacorilant 150 mg once daily (QD)
- Nab-paclitaxel 100 mg/m^2 (Active Comparator): Patients receive nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Nab-paclitaxel 100 mg/m^2

INTERVENTIONS:
Drug: Nab-paclitaxel 80 mg/m^2 — Nab-paclitaxel is administered as intravenous (IV) infusion over 30-40 minutes on Days 1, 8, and 15 of each 28-day cycle.
  Arms: Nab-paclitaxel 80 mg/m^2 with Relacorilant 150 mg
Drug: Relacorilant 150 mg once daily (QD) — Relacorilant is administered as capsules for oral dosing.
  Arms: Nab-paclitaxel 80 mg/m^2 with Relacorilant 150 mg
Drug: Nab-paclitaxel 100 mg/m^2 — Nab-paclitaxel is administered as IV infusion on Day 1, 8, and 15 of each 28-day cycle.
  Arms: Nab-paclitaxel 100 mg/m^2

SUMMARY:
The primary objectives of this study are to evaluate progression-free survival (PFS) by blinded independent central review (BICR) and overall survival (OS) (evaluated independently, as dual primary endpoints) in patients treated with intermittent regimen of Relacorilant in combination with nab-paclitaxel compared with patients treated with nab-paclitaxel monotherapy.

DETAILED DESCRIPTION:
As there are no currently approved therapies or effective standard of care for heavily pretreated patients with ovarian cancer who have exhausted single-agent chemotherapy and/or bevacizumab, the combination of intermittently administered relacorilant and nab-paclitaxel may demonstrate a substantial improvement without increased toxicity compared with nab-paclitaxel.

Patients will receive study treatment until confirmed progressive disease (PD) or unacceptable toxicity. All patients will be followed for the collection of study endpoints, inclusive of disease progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Institutional Review Board/Independent Ethics Committee-approved informed consent form prior to study-specific screening procedures.
* Confirmed histologic diagnosis of high-grade (Grade 3) serous, epithelial ovarian, primary peritoneal, or fallopian tube carcinoma.
* Patients must have platinum-resistant disease (defined as RECIST v1.1 defined progression <6 months from completion of a platinum-containing therapy).
* Must consent to provide archival tumor-tissue block or slides. Patients may consent to an optional tumor biopsy if archival tumor is unavailable.
* Has a life expectancy of ≥3 months.
* At least one lesion that meets the definition of measurable disease by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Able to comply with protocol requirements.
* Able to swallow and retain oral medication and does not have uncontrolled emesis.
* Received at least 1 but ≤3 lines of prior systemic anticancer therapy and at least 1 prior line of platinum therapy and prior treatment with bevacizumab is required.
* Has adequate organ function meeting the following laboratory-test criteria: Absolute neutrophil count (ANC) ≥1500 cells/mm^3, Platelet count ≥100,000/mm^3, Hemoglobin ≥9 g/dL, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN), or ≤5 × ULN in context of liver metastases, Total bilirubin ≤1.5 × ULN, and Albumin ≥3 g/dL, and creatinine clearance >40 mL/min/1.73 m^2 (measured or estimated).
* Negative pregnancy test for patients of childbearing potential; patients of childbearing potential must agree to use highly effective contraceptive method(s); hormonal contraceptives are not allowed.
* Coronavirus disease (COVID-19) approved vaccines are accepted concomitant medications when recommended by the Investigator.

Exclusion Criteria:

* Has clinically relevant toxicity from prior systemic anticancer therapies or radiotherapy that has not resolved to ≤Grade 1 prior to randomization.
* Has had any major surgery within 4 weeks prior to randomization.
* Has low-grade endometrioid, clear cell, mucinous, or sarcomatous histology, or mixed tumors containing any of these histologies, or low-grade or borderline ovarian tumor.
* Has primary platinum-refractory disease, defined as disease that did not respond to or has progressed ≤1 month of the last dose of first-line platinum-containing chemotherapy.
* Has not received prior bevacizumab treatment.
* Has been treated with the following prior to randomization: chemotherapy, immunotherapy, investigational agent treatments for disease under study within 28 days before first dose of study drug, radiotherapy not completed at least 2 weeks prior to first dose of study drug, hormonal anticancer therapies within 7 days of first dose of study drug, and systemic, inhaled, or prescription strength topical corticosteroids within 21 days of first dose of study drug.
* Has received wide-field radiation to more than 25% of marrow-bearing areas.
* Has toxicities of prior therapies that have not resolved the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, ≤Grade 1.
* Requires treatment with chronic or frequently used oral corticosteroids for medical conditions or illnesses.
* Has a history of severe hypersensitivity or severe reaction to any of the study drugs.
* Is receiving concurrent treatment with mifepristone or other glucocorticoid receptor (GR) modulators.
* Has peripheral neuropathy from any cause >Grade 1.
* Pregnant or lactating patients or patients expecting to conceive children within the projected duration of the trial, starting with the screening visit through at least 1 month after the last dose of relacorilant, or 6 months after the last dose of nab-paclitaxel whichever is the longest.
* Has clinically significant uncontrolled condition(s) or condition which, in the opinion of the Investigator, may confound the results of the trial or interfere with the patient's safety or participation.
* Has current chronic/active infection with human immunodeficiency virus or current chronic/active infection with hepatitis C virus or hepatitis B virus.
* Has any untreated or symptomatic central nervous system (CNS) metastases.
* Patients with a history of other malignancy within 3 years prior to randomization
* Is taking a concomitant medication that is a strong cytochrome P450 (CYP)3A inhibitor or strong CYP3A inducer, or that is a substrate of CYP3A with a narrow therapeutic window.
* Concurrent treatment on other investigational treatment studies for the treatment of ovarian, fallopian tube, or primary peritoneal cancer.
* Has received a live vaccine within 30 days of prior to the study start date.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival as Assessed by BICR | Up to 24 months from enrollment of the last patient
  Time from randomization until the time of first documented progressive disease (PD) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death due to any cause, whichever occurs first
Overall survival | Up to 24 months from enrollment of the last patient
  Time from randomization to death by any cause

SECONDARY OUTCOMES:
PFS as Assessed by the Investigator | Up to 24 months from enrollment of the last patient
  Time from randomization until the time of first documented progressive disease (PD) by RECIST v1.1, or death due to any cause, whichever occurs first
Objective Response as Assessed by BICR | Up to 24 months from enrollment of the last patient
  Proportion of patients with measurable disease at baseline who attain CR or PR by RECIST v1.1.
Best Overall Response as Assessed by BICR | Up to 24 months from enrollment of the last patient
  Proportion of patients with measurable disease at baseline who attain CR or PR as best response by RECIST v1.1.
Duration of Response as Assessed by BICR | Up to 24 months from enrollment of the last patient
  Time from when response (CR or PR per RECIST v1.1) is first documented to first objectively documented PD or death (whichever occurs first)
Clinical benefit rate as assessed by BICR | 24 weeks
  Proportion of patients who attain CR, PR, or stable disease (SD) per RECIST v1.1.
Cancer Antigen (CA)-125 Response | Up to 24 months from enrollment of the last patient
  Cancer antigen (CA)-125 response will be assessed per Gynecologic Cancer Intergroup (GCIG) criteria defined as ≥50% reduction in CA-125 from a pre-treatment sample and maintained for ≥28 days in patients with a pretreatment sample that is at least twice the upper limit of the reference range within 2 weeks before starting the treatment. In addition, patients who have a CA-125 response and whose CA-125 level falls to within the reference range will be classified as CA-125 complete responders.
Combined Response According to RECIST v1.1 and GCIG Criteria | Up to 24 months from enrollment of the last patient
  Combined response will be assessed for PD per RECIST v1.1 and for CA-125 response per GCIG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Pai, MD, Study Director — Corcept Therapeutics
Locations (117):
- United States (44):
  - Site 318, Phoenix, Arizona
  - Site 277, Tucson, Arizona
  - Site 350, Irvine, California
  - Site 364, La Jolla, California
  - Site 150, Palo Alto, California
  - Site 278, San Francisco, California
  - Site 014, San Francisco, California
  - Site 316, Solvang, California
  - Site 032, Aurora, Colorado
  - Site 335, Miami Beach, Florida
  - Site 042, Weston, Florida
  - Site 009, Atlanta, Georgia
  - Site 272, Atlanta, Georgia
  - Site 372, Gainesville, Georgia
  - Site 291, Savannah, Georgia
  - Site 315, Evanston, Illinois
  - Site 314, Hinsdale, Illinois
  - Site 346, Urbana, Illinois
  - Site 339, Indianapolis, Indiana
  - Site 200, Overland Park, Kansas
  - Site 334, Overland Park, Kansas
  - Site 279, Louisville, Kentucky
  - Site 128, Boston, Massachusetts
  - Site 288, New Brunswick, New Jersey
  - Site 292, Albuquerque, New Mexico
  - Site 275, Flushing, New York
  - Site 298, Cincinnati, Ohio
  - Site 304, Cincinnati, Ohio
  - Site 280, Portland, Oregon
  - Site 317, Portland, Oregon
  - Site 049, Portland, Oregon
  - Site 337, Bethlehem, Pennsylvania
  - Site 127, Pittsburgh, Pennsylvania
  - Site 276, Rapid City, South Dakota
  - Site 368, Germantown, Tennessee
  - Site 281, Nashville, Tennessee
  - Site 229, Austin, Texas
  - Site 312, Bedford, Texas
  - Site 297, Fort Worth, Texas
  - Site 392, San Antonio, Texas
  - Site 301, The Woodlands, Texas
  - Site 300, Norfolk, Virginia
  - Site 365, Richmond, Virginia
  - Site 121, Milwaukee, Wisconsin
- Argentina (8):
  - Site 393, CABA, Buenos Aires
  - Site 381, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Site 415, Córdoba, Córdoba Province
  - Site 401, Córdoba, Córdoba Province
  - Site 395, Córdoba, Córdoba Province
  - Site 404, Mendoza, Mendoza Province
  - Site 391, Rosario, Santa Fe Province
  - Site 412, Rosario, Santa Fe Province
- Australia (4):
  - Site 426, St Leonards, New South Wales
  - Site 417, Benowa, Queensland
  - Site 414, Melbourne, Victoria
  - Site 419, Melbourne, Victoria
- Belgium (6):
  - Site 328, Aalst
  - Site 109, Brussels
  - Site 326, Charleroi
  - Site 325, Hasselt
  - Site 108, Leuven
  - Site 327, Liège
- Brazil (13):
  - Site 424, Brasília, Brasília - DF
  - Site 382, Fortaleza, Ceará
  - Site 384, Salvador, Estado de Bahia
  - Site 383, Belo Horizonte, Minas Gerais
  - Site 390, Natal, Rio Grande do Norte
  - Site 413, São Paulo, São Paulo
  - Site 421, Porto Alegre
  - Site 380, Rio de Janeiro
  - Site 376, São Paulo
  - Site 389, São Paulo
  - Site 413, São Paulo
  - Site 374, São Paulo
  - Site 001, São Paulo
- Canada (2):
  - Site 117, Toronto, Ontario
  - Site 273, Montreal, Quebec
- France (6):
  - Site 306, Lille
  - Site 347, Montpellier
  - Site 307, Nancy
  - Site 310, Nice
  - Site 289, Paris
  - Site 323, Plérin
- Hungary (3):
  - Site 322, Budapest
  - Site 290, Debrecen
  - Site 348, Győr
- Israel (3):
  - Site 309, Haifa
  - Site 080, Jerusalem
  - Site 203, Tel Aviv
- Italy (8):
  - Site 321, Catania
  - Site 320, Legnago
  - Site 122, Milan
  - Site 295, Pavia
  - Site 161, Roma
  - Site 124, Rome
  - Site 293, Torino
  - Site 319, Treviso
- Poland (3):
  - Site 341, Gdynia
  - Site 331, Poznan
  - Site 329, Siedlce
- South Korea (8):
  - Site 397, Gyeonggi-do
  - Site 399, Seoul
  - Site 398, Seoul
  - Site 403, Seoul
  - Site 400, Seoul
  - Site 396, Seoul
  - Site 402, Seoul
  - Site 409, Seoul
- Spain (3):
  - Site 349, Badalona
  - Site 311, San Sebastián
  - Site 330, Valencia
- United Kingdom (6):
  - Site 367, Brighton, East Sussex
  - Site 351, Taunton, Somerset
  - Site 366, Cheltenham
  - Site 055, London
  - Site 344, Manchester
  - Site 345, Northwood

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olawaiye AB, Gladieff L, O'Malley DM, Kim JW, Garbaos G, Salutari V, Gilbert L, Mileshkin L, Devaux A, Hopp E, Lee YJ, Oaknin A, Scaranti M, Kim BG, Colombo N, McCollum ME, Diakos C, Clamp A, Leiser AL, Balazs B, Monk BJ, Scandurra G, McClung E, Kaczmarek E, Slomovitz B, De La Cueva H, de Carvalho Calabrich AF, Cassani C, You B, Van Gorp T, Churruca C, Caruso G, Nicum S, Bagameri A, Artioli G, Bodnar L, Kang S, Vergote I, Kesner-Hays A, Pashova HI, Pai SG, Tudor IC, Jubb AM, Lorusso D. Relacorilant and nab-paclitaxel in patients with platinum-resistant ovarian cancer (ROSELLA): an open-label, randomised, controlled, phase 3 trial. Lancet. 2025 Jun 21;405(10496):2205-2216. doi: 10.1016/S0140-6736(25)01040-2. Epub 2025 Jun 2. PMID 40473448
- [Derived] Olawaiye AB, Kim JW, Bagameri A, Bishop E, Chudecka-Glaz A, Devaux A, Gladieff L, Gordinier ME, Korach J, McCollum ME, Mileshkin L, Monk BJ, Nicum S, Nogueira-Rodrigues A, Oaknin A, O'Malley DM, Orlando M, Dreiling L, Tudor IC, Lorusso D. Clinical Trial Protocol for ROSELLA: a phase 3 study of relacorilant in combination with nab-paclitaxel versus nab-paclitaxel monotherapy in advanced platinum-resistant ovarian cancer. J Gynecol Oncol. 2024 Jul;35(4):e111. doi: 10.3802/jgo.2024.35.e111. PMID 39032926
- [Derived] Colombo N, Van Gorp T, Matulonis UA, Oaknin A, Grisham RN, Fleming GF, Olawaiye AB, Nguyen DD, Greenstein AE, Custodio JM, Pashova HI, Tudor IC, Lorusso D. Relacorilant + Nab-Paclitaxel in Patients With Recurrent, Platinum-Resistant Ovarian Cancer: A Three-Arm, Randomized, Controlled, Open-Label Phase II Study. J Clin Oncol. 2023 Oct 20;41(30):4779-4789. doi: 10.1200/JCO.22.02624. Epub 2023 Jun 26. PMID 37364223